CLINICAL TRIAL: NCT02294292
Title: Therapeutic Approach to Diastolic Dysfunction in Chronic Liver Disease Patients and Its' Impact on Morbidity and Mortality
Brief Title: Therapeutic Approach to Diastolic Dysfunction in Chronic Liver Disease Patients and Its Impact on Morbidity and Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-CLD-DD-01
Record Dates: First submitted 2014-06-09; First posted 2014-11-19 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2016-02

CONDITIONS: Diastolic Dysfunction; Chronic Liver Disease
MeSH Terms: interventions — Carvedilol; Ivabradine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol + Ivabradine (Experimental): Carvedilol started to achieve target HR (heart rate) reduction to 60/min, to a lowest permissible 50-55/ min ; provided Systolic Blood Pressure> 90 mmHg.
  if carvedilol is not tolerated,Ivabradine is added in a dose starting 2.5 mg BD to a maximum of 15 mg/day to ensure targeted heart rate reduction
  Interventions: Drug: Carvedilol; Drug: Ivabradine
- Endoscopic Variceal Ligation (EVL) (Active Comparator)
  Interventions: Procedure: Endoscopic Variceal Ligation

INTERVENTIONS:
Drug: Carvedilol — Carvedilol started to achieve target HR (heart rate) reduction to 60/min, to a lowest permissible 50-55/ min ; provided Systolic Blood Pressure> 90 mmHg.
  Arms: Carvedilol + Ivabradine
Drug: Ivabradine — Carvedilol started to achieve target HR (heart rate) reduction to 60/min, to a lowest permissible 50-55/ min ; provided Systolic Blood Pressure> 90 mmHg.
  If carvedilol is not tolerated,Ivabradine is added in a dose starting 2.5 mg BD to a maximum of 15 mg/day to ensure targeted heart rate reduction
  Arms: Carvedilol + Ivabradine
Procedure: Endoscopic Variceal Ligation
  Arms: Endoscopic Variceal Ligation (EVL)

SUMMARY:
Cirrhotic cardiomyopathy is defined as a chronic cardiac dysfunction in patients with cirrhosis. It is suspected that this specific cardiac dysfunction contributes to the onset of complications in liver disease. The purpose of this prospective, randomized controlled trial is to determine whether carvedilol can revert cardiac dysfunction i.e. left ventricular diastolic dysfunction secondary to cirrhosis, and prevent complications (renal dysfunction, worsening cardiac function, and mortality).

ELIGIBILITY:
Inclusion Criteria:

Patients with cirrhosis who have been diagnosed by clinical, biochemical,or histological (when available) criteria plus ultrasound imaging.

* Age range of 18-60 years
* Cirrhosis as diagnosed by histology or clinical, laboratory and USG (UltraSonography) findings,
* Upper GI bleed who are undergoing secondary endoscopic variceal ligation for eradication of varices

Exclusion Criteria:

* Age >60 years
* Chronic renal disease
* Pregnancy and peripartum cardiomyopathy
* Hypertension
* Coronary artery disease
* Valvular heart disease
* Sick sinus syndrome/ Pacemaker
* Cardiac rhythm disorder
* Hypothyroidism
* Hyperthyroidism
* Portal vein thrombosis
* Transjugular intrahepatic porto systemic shunt (TIPS) insertion
* Hepatocellular carcinoma
* Anemia Hb < 8gm/dl in females, and < 9 gm/dl in males

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Progression of cirrhosis and its complications. | 1 Year

SECONDARY OUTCOMES:
Improvement in left ventricular diastolic function in either arm. | 1 Year
Renal function | 1 Year
  Renal function is being checked- urea, creatinine, urine sediment, and creatinine clearance as calculated by Cockcroft - Gault formula
Serum level of Brain Natriuretic Peptide. | 1 Year
Mortality | 1 Year
Quality of life | 1 Year
Electrophysiologic modifications | 1 Year
  Electrophysiological changes checked are QTc interval, documentation of arrhythmias
Serum level of catecholamines | 1 year
Serum level of plasma renin activity | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Premkumar M, Rangegowda D, Vyas T, Khumuckham JS, Shasthry SM, Thomas SS, Goyal R, Kumar G, Sarin SK. Carvedilol Combined With Ivabradine Improves Left Ventricular Diastolic Dysfunction, Clinical Progression, and Survival in Cirrhosis. J Clin Gastroenterol. 2020 Jul;54(6):561-568. doi: 10.1097/MCG.0000000000001219. PMID 31305281